CLINICAL TRIAL: NCT04426279
Title: Morbimortality of Covid-19 in Patients With Chronic Inflammatory Rheumatism Treated With Immunosuppressants
Acronym: CORhum
Status: Terminated | Type: Observational
Why Stopped: Number of patients not reached during the inclusion period, end of funding.
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_49; 2020-A01650-39 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-01

CONDITIONS: Sars-CoV2; Rheumatoid Arthritis; Rheumatic Diseases
Keywords: Immunotherapy; chronic inflammatory rheumatism
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with chronic inflammatory rheumatism
  Interventions: Other: questionnaire assesment

INTERVENTIONS:
Other: questionnaire assesment — 15-minute face-to-face questionnaire

SUMMARY:
A retrospective monocentric study with large active files of patients monitored for rheumatoid arthritis, spondyloarthritis and systemic lupus erythematosus with as main endpoint the morbimortality of Covid-19 in these patients (number of patients hospitalized in conventional units and/or in intensive care and/or deceased). The results will be compared with those of the general population based on the epidemiological data of Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis on conventional synthetic DMARD (csDMARDs) +/- biological DMARD (bDMARDs) or targeted synthetic DMARD (tsDMARDs) +/- corticosteroid therapy meeting ACR/EULAR 2010 classification criteria
* Patients with spondylarthritison biological DMARD or targeted synthetic DMARD +/- conventional synthetic DMARD +/- non-steroidal anti-inflammatory drugs meeting ASAS classification criteria
* Patients with systemic lupus erythematosus on hydroxychloroquine +/- conventional synthetic DMARD +/- corticosteroid therapy +/- biological DMARD meeting ACR/EULAR 2019 classification criteria

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammatory rheumatic diseases who are immunosuppressed: rheumatoid arthritis/spondylarthritis [individualized psoriatic spondyloarthritis and rheumatism]/systemic lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
analysis of Covid-19-related morbidity and mortality in patients with IRC under IS. | At 6 months
  the number of patients with severe Covid-19 who were admitted to a conventional unit and/or an ICU and/or deceased, during the Covid-19 epidemic wave (from March to August 2020) among patients with IRC under IS. The diagnosis of Covid-19 is either confirmed by diagnostic test (RT-PCR), or by a physician, or by serology. The results will be compared with those of the general population based on Covid-19 epidemiological data.

SECONDARY OUTCOMES:
To evaluate the frequency of Covid-19 in patients with IRC under IS. | At 6 months
  Diagnosis of Covid-19 either confirmed by diagnostic test (RT-PCR), or by a physician, or by serology.
To compare the morbidity and mortality of patients with IRC under IS during the Covid-19 epidemic wave (March to August 2020) with the six months prior to this wave (September 2019 to February 2020). | At 6 months
  The number of patients admitted to conventional unit and/or ICU and/or deceased among patients with IRC under IS between the Covid-19 epidemic wave (March to August 2020) and the six-month period preceding it (September to February 2020).
Patients' conduct in relation to their treatment during the epidemic wave (maintenance, modification or discontinuation) and the impact on their disease (loss of remission, flare, corticosteroids requirement and need for switch of DMARD therapy) | At 6 months
  The number of patients who maintained, modified, or discontinued their treatment. Treatment modification will be assessed by the number of weeks of treatment not taken, the number of injections not given, the number of delayed or missed infusions. Among those who have modified or stopped their treatment, the impact on their diseases will be evaluated by the loss of remission, the patient's opinion on the notion of relapse, the increase or initiation of corticosteroid therapy and the substantive change in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Guillaume Letarouilly, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Monti S, Balduzzi S, Delvino P, Bellis E, Quadrelli VS, Montecucco C. Clinical course of COVID-19 in a series of patients with chronic arthritis treated with immunosuppressive targeted therapies. Ann Rheum Dis. 2020 May;79(5):667-668. doi: 10.1136/annrheumdis-2020-217424. Epub 2020 Apr 2. No abstract available. PMID 32241793
- [Background] Gianfrancesco MA, Hyrich KL, Gossec L, Strangfeld A, Carmona L, Mateus EF, Sufka P, Grainger R, Wallace Z, Bhana S, Sirotich E, Liew J, Hausmann JS, Costello W, Robinson P, Machado PM, Yazdany J; COVID-19 Global Rheumatology Alliance Steering Committee. Rheumatic disease and COVID-19: initial data from the COVID-19 Global Rheumatology Alliance provider registries. Lancet Rheumatol. 2020 May;2(5):e250-e253. doi: 10.1016/S2665-9913(20)30095-3. Epub 2020 Apr 16. No abstract available. PMID 32309814
- [Background] Haberman R, Axelrad J, Chen A, Castillo R, Yan D, Izmirly P, Neimann A, Adhikari S, Hudesman D, Scher JU. Covid-19 in Immune-Mediated Inflammatory Diseases - Case Series from New York. N Engl J Med. 2020 Jul 2;383(1):85-88. doi: 10.1056/NEJMc2009567. Epub 2020 Apr 29. No abstract available. PMID 32348641
- [Background] Michaud K, Wipfler K, Shaw Y, Simon TA, Cornish A, England BR, Ogdie A, Katz P. Experiences of Patients With Rheumatic Diseases in the United States During Early Days of the COVID-19 Pandemic. ACR Open Rheumatol. 2020 Jun;2(6):335-343. doi: 10.1002/acr2.11148. Epub 2020 May 9. PMID 32311836
- [Background] Favalli EG, Ingegnoli F, De Lucia O, Cincinelli G, Cimaz R, Caporali R. COVID-19 infection and rheumatoid arthritis: Faraway, so close! Autoimmun Rev. 2020 May;19(5):102523. doi: 10.1016/j.autrev.2020.102523. Epub 2020 Mar 20. PMID 32205186